CLINICAL TRIAL: NCT06961929
Title: IEEM-Heat and Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU20250699
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Hyperthermia
Keywords: heat wave; cardiovascular; cooling strategies; myocardial perfusion
MeSH Terms: conditions — Heart Failure; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Congestive Heart Failure (CHF) (Active Comparator)
  Interventions: Other: Control Trial; Other: Water-saturated T-shirt trial; Other: Skin-Wetting Trial
- Individuals without Congestive Heart Failure (Control) (Active Comparator)
  Interventions: Other: Control Trial; Other: Water-saturated T-shirt trial; Other: Skin-Wetting Trial

INTERVENTIONS:
Other: Control Trial — All participants will be exposed to a period of hyperthermia (hot and dry). In this condition, participants will not be given an experimental cooling modality.
Other: Water-saturated T-shirt trial — All participants will be exposed to a period of hyperthermia (hot and dry). In this condition, participants will also wear a T-shirt that has been saturated with water.
Other: Skin-Wetting Trial — All participants will be exposed to a period of hyperthermia (hot and dry). In this condition, participants will also be sprayed with water periodically.

SUMMARY:
We will test the hypothesis that increasing skin wetness, and thus evaporative cooling, will attenuate the increase in core body temperature and accompanying cardiac stress during heat wave conditions in individuals with congestive heart failure. Secondly, we propose that wearing a water-saturated T-shirt will also be beneficial to attenuate the increase in core body temperature and accompanying cardiac stress during heat wave conditions in individuals with congestive heart failure. To accomplish these objectives, individuals with congestive heart failure and otherwise healthy control individuals will be exposed to the simulated heat wave condition (hot and dry) with the following cooling modalities: A) control trial (no limb immersion or skin wetting), B) skin wetting only trial, and C) water-saturated T-shirt trial in a randomized crossover fashion. Thermoregulatory and cardiovascular responses will be evaluated throughout these simulated heat wave exposures.

Primary outcomes variables will be skin and core temperatures, while secondary variables will include measures of cardiovascular stress, myocardial perfusion, heart rate, and echo-based measures of cardiac function.

ELIGIBILITY:
Inclusion Criteria for healthy control participants:

* Participants must be free of any significant underlying medical problems based upon a detailed medical history and physical exam, and normal resting electrocardiogram. Participants must be 35+ years.

Exclusion Criteria for healthy control participants:

* Known heart disease; other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, lung disease, etc.; as well as serious abnormalities detected on routine screening. Current smokers, as well as individuals who regularly smoked within the past 12 months, will be excluded. Subjects who cannot be age and gender matched to an individual in the heart failure group will be excluded.

Inclusion Criteria for Participants with CHF:

- The participant must have a diagnosis of congestive heart failure (e.g., heart failure with reduced ejection fraction), with the severity categorized as New York Heart Association (NYHA) class II or III. Participants must be 35+ years.

Exclusion Criteria for Participants with CHF:

-Patients who do not have confirmed diagnosis of NYHA class II or III heart failure will be excluded from the clinical group. Potential participants with cancer, diabetes, neurological disease, lung disease, and/or uncontrolled hypertension will be excluded. Potential participants with a left bundle branch block on ECG will be excluded. Patients on anticoagulant therapy will also be excluded. Current smokers, as well as individuals who regularly smoked within the past 12 months, will be excluded. Further exclusions will include severe valvular or congenital heart disease, acute myocarditis, NYHA Class IV heart failure, and/or manifest/provocable ischemic heart disease.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Core Body Temperature while wearing a water-saturated T-shirt | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Core body temperature will be measured from gastrointestinal temperature via an ingestible telemetric pill or rectal temperature via telemetric pill suppository or rectal thermistor. Core body temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in core body temperature.
Change in Core Body Temperature in Skin-Wetting Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Core body temperature will be measured from gastrointestinal temperature via an ingestible telemetric pill or rectal temperature via telemetric pill suppository or rectal thermistor. Core body temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in core body temperature.
Change in Core Body Temperature in Control Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Core body temperature will be measured from gastrointestinal temperature via an ingestible telemetric pill or rectal temperature via telemetric pill suppository or rectal thermistor. Core body temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in core body temperature.
Change in Skin Temperature in while wearing a water-saturated T-shirt | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin. Skin temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in skin temperature.
Change in Skin Temperature in Skin-Wetting Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin. Skin temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in skin temperature.
Change in Skin Temperature in Control Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin. Skin temperature will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those temperatures will reflect the change in skin temperature.

SECONDARY OUTCOMES:
Change in Heart Rate while wearing a water-saturated T-shirt | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Heart rate will be measured from ECG electrodes attached to the participant. Heart rate will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in heart rate.
Change in Heart Rate in Skin-Wetting Trial | Prior to and after each simulated heat wave exposure (approximately 210minutes.)
  Heart rate will be measured from ECG electrodes attached to the participant. Heart rate will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in heart rate.
Change in Heart Rate in Control Trial | Prior to and after each simulated heat wave exposure (approximately 210minutes.)
  Heart rate will be measured from ECG electrodes attached to the participant. Heart rate will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in heart rate.
Rate Pressure Product while wearing a water-saturated T-shirt | At the end of each heat wave exposure. Approximately 210minutes after the start of the heat wave simulation.
  Rate Pressure Product is calculated by multiplying Systolic Blood Pressure and Heart Rate.
Rate Pressure Product in Skin-Wetting Trial | At the end of each heat wave exposure. Approximately 210minutes after the start of the heat wave simulation.
  Rate Pressure Product is calculated by multiplying Systolic Blood Pressure and Heart Rate.
Rate Pressure Product in Control Trial | At the end of each heat wave exposure. Approximately 210minutes after the start of the heat wave simulation.
  Rate Pressure Product is calculated by multiplying Systolic Blood Pressure and Heart Rate.
Change in Cardiac Output while wearing a water-saturated T-shirt | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Cardiac output (how much blood is ejected from the heart) will be measured using echocardiography. Cardiac output will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in cardiac output.
Change in Cardiac Output in Skin-Wetting Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Cardiac output (how much blood is ejected from the heart) will be measured using echocardiography. Cardiac output will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in cardiac output.
Cardiac Output in Control Trial | Prior to and after each simulated heat wave exposure (approximately 210 minutes.)
  Cardiac output (how much blood is ejected from the heart) will be measured using echocardiography. Cardiac output will be measured at baseline as well as at the end of the hyperthermia simulation. The difference of those heart rates will reflect the change in cardiac output.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Exercise and Environmental Medicine - Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No